CLINICAL TRIAL: NCT03157973
Title: Modern Technology For Learning and Psychosocial Support In Patients With Abdominal Aortic Aneurysm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Olga Nilsson, RN, SC, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnr 2016/1253-31/4
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Aortic Aneurysm
Keywords: Information Literacy; Nursing Care; Social Support
MeSH Terms: conditions — Aortic Aneurysm | interventions — Early Intervention, Educational

STUDY DESIGN:
Masking Description: The nature of the intervention rules out masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education intervention (Experimental)
  Interventions: Other: Education intervention
- Standard of Care (No Intervention)

INTERVENTIONS:
Other: Education intervention — eHealth tool and standardized nurse-led follow-up.
  Arms: Education intervention

SUMMARY:
This study evaluates the effects of an eHealth tool and psychosocial support on anxiety, depression and health-related quality of life in patients undergoing surgical treatment for abdominal aortic aneurysm (AAA). Participants in the intervention group will receive access to the eHealth tool and structured follow-up with a contact nurse, the control group will receive standard of care.

DETAILED DESCRIPTION:
Abdominal aortic anuerysm (AAA) is associated with a decreased health-related quality of life (HRQoL) both at diagnosis and during surgical treatment, although recent studies report somewhat contradictory results. In qualitative research, it has been shown that the health care system fails to meet the patients' information need, as well as their need for psychosocial support during the care process. The aim of this study is therefore to evaluate the effects of an intervention comprising an eHealth tool with individualized information in combination with structured follow-up with a contact nurse on anxiety, depression and HRQoL in patients undergoing surgical treatment for AAA.

Patients who are planned for elective surgical treatment, fulfil the inclusion criteria and none of the exclusion criteria will fill out questionnaires. The control group will receive information and follow-up per institution's standard of care. The intervention group will be given access to the eHealth tool, containing individualized information about the condition, surgical procedure and self-care. They will also receive structured follow-up by a contact nurse at discharge, 3 and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak and understand Swedish
* Planned for elective surgical repair of an abdominal aortic aneurysm

Exclusion Criteria:

* Severe visual impairment or blindness
* Severe hearing impairment or deafness
* Diagnosed dementia
* Medical condition with a suspected life expectancy of < 1 year.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 12 months
  A validated self-assessment scale that measures symptoms of anxiety and depression in a non-psychiatric population.

SECONDARY OUTCOMES:
SF12 | 12 months
  A 12-item questionnaire that measures 8 dimensions of physical and mental health.
Quality from the patient's perspective (QPP) | 12 months
  A validated self-assessment scale measuring patient perceived quality of care.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecka Hultgren, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Vascular Surgery, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson O, Stenman M, Letterstal A, Hultgren R. One-year results of an eHealth intervention on anxiety in patients undergoing abdominal aortic aneurysm surgery: randomized clinical trial. BJS Open. 2024 Dec 30;9(1):zrae144. doi: 10.1093/bjsopen/zrae144. PMID 39812416
- [Derived] Nilsson O, Stenman M, Letterstal A, Hultgren R. A randomized clinical trial of an eHealth intervention on anxiety in patients undergoing abdominal aortic aneurysm surgery. Br J Surg. 2021 Aug 19;108(8):917-924. doi: 10.1093/bjs/znab151. PMID 34021309